CLINICAL TRIAL: NCT00746694
Title: Epidemiological Study to Assess the Management of Palmar-plantar Erythrodysesthesia (PPE) in Patients With Metastatic Ovarian or Breast Cancer Treated With Pegylated Liposomal Doxorubicin
Brief Title: A Study to Determine the Management of Palmar-plantar Erythrodysesthesia (PPE) in Patients With Metastatic Ovarian or Breast Cancer Treated With Caelyx (Study P05020)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05020
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2011-01-17 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Ovarian Neoplasms; Breast Neoplasms; Paresthesia
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Paresthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Caelyx: Participants with metastatic breast or ovarian cancer treated with Caelyx as part of standard treatment and according to data sheet approved indications.

SUMMARY:
The objective of this trial is to study the management of PPE in participants with metastatic ovarian or breast cancer treated with Caelyx, and determine the frequency of use of pharmacological treatment (preventive or therapeutic) for PPE and compliance of educational recommendations for PPE.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older.
* Participants with metastatic breast or ovarian cancer who are receiving treatment with pegylated liposomal doxorubicin.
* Participants who have given their written consent.

Exclusion Criteria:

* Participants who are currently participating in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic ovarian or breast cancer, to be recruited from the Oncology Departments of 16 centers for a period of 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Caelyx: Caelyx, 2mg/ml concentrate for solution for intravenous (IV) administration. 50mg/m2 IV once every 4 weeks. Participants with metastatic breast or ovarian cancer treated with Caelyx as part of standard treatment.
Period: Overall Study
Arm/Group | Caelyx
Started | 154
Completed | 154
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Caelyx
Number analyzed (Participants) | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 154

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Concomitant Treatment Strategies to Manage Palmar-Plantar Erythrodysesthesia (PPE)
Description: Participants treated with Caelyx who developed PPE and the categories of specific treatment strategies that were prescribed to manage the symptoms of PPE.
  Participants counted under the strategies: Keep Skin Hydrated; Avoid Sweating and Physical Activity; Avoid Tight-Fitting Clothing; Local Cooling of Hands and Feet; were those who either always or sometimes followed it.
Time Frame: Participants will do a single visit, but cases will be collected during a period of 12 months.
Measure: Number; unit: Participants
Arm/Group | Caelyx
Number analyzed (Participants) | 154
Participants
  Oral Dexamethosone | 10
  Pyridoxine | 8
  Topical Corticosteroids | 8
  Topical Dimethyl Sulfoxide | 3
  Intravenous Dexamethasone | 1
  Prostaglandins | 1
  Avoid Excessive Heat/Water | 14
  Keep Skin Hydrated | 14
  Avoid Sweating and Physical Activity | 14
  Avoid Tight-Fitting Clothing | 14
  Local Cooling of Hands and Feet | 13

2. Primary Outcome: Number of Participants That Received Curative Treatment and/or Prophylaxis Treatment for PPE
Description: The number of participants who were treated with Caelyx, and who received either prophylactic treatment alone, or curative treatment alone, or both prophylactic and curative treatment for PPE.
Time Frame: Participants will do a single visit, but cases will be collected during a period of 12 months.
Measure: Number; unit: Participants
Arm/Group | Caelyx
Number analyzed (Participants) | 154
Participants
  Curative Treatment | 14
  Prophylaxis | 52
  Curative & Prophylactic Treatment | 6

ADVERSE EVENTS:
Arm/Group | Caelyx
Serious Adverse Events (participants affected / at risk) | 3/154
Other Adverse Events (participants affected / at risk) | 122/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx (N=154)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx (N=154)
Neutropenia (Blood and lymphatic system disorders) | 18 (18)
Abdominal pain (Gastrointestinal disorders) | 11 (11)
Constipation (Gastrointestinal disorders) | 21 (21)
Diarrhoea (Gastrointestinal disorders) | 21 (21)
Nausea (Gastrointestinal disorders) | 51 (51)
Stomatitis (Gastrointestinal disorders) | 68 (68)
Vomiting (Gastrointestinal disorders) | 15 (15)
Asthenia (General disorders) | 61 (61)
Anorexia (Metabolism and nutrition disorders) | 27 (27)
Alopecia (Skin and subcutaneous tissue disorders) | 44 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study data may be used in general publications or at conferences. Authorship will be attributed to those responsible for preparing the report and/or those who had a relevant part in designing the study. Whenever publication rules allow, all investigators will be listed individually.

Investigators may publish their data individually. In this case investigators will notify the study sponsor, including the communication/manuscript to be published, at least 30 days before submission.